CLINICAL TRIAL: NCT05232331
Title: Effect of Nitrate-rich Vegetable Intake on Inflammatory Molecule Levels, Nitrate-reducing Capacity and Oral Microbiota Composition in Patients With Periodontitis
Brief Title: Intake of Nitrate-rich Vegetables and Their Effect on Inflammatory Molecules and Oral Microbiota of Patients With Periodontitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-02721
Record Dates: First submitted 2021-11-26; First posted 2022-02-09 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Periodontal Diseases; Periodontitis
Keywords: Nitrates; Vegetables; Oral Microbiota; Periodontitis; Inflammatory molecules
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Single blind. Dentists in charge of assessing dental clinical parameters, as well as researchers performing the analysis of the oral microbiota, will be unaware of the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This group will receive non-surgical periodontal treatment, however they will not receive any modification to their diet
- Intervention (Experimental): This group will receive non-surgical periodontal treatment, and also as a treatment of interest, will receive the indication to consume ~ 350 mg of nitrate from vegetables, as well as an accompaniment to achieve this objective.
  Interventions: Dietary Supplement: Intake of nitrate rich vegetables

INTERVENTIONS:
Dietary Supplement: Intake of nitrate rich vegetables — Nutritional intervention for 10 weeks to increase the consumption of vegetables rich in nitrate. At the beginning of the NSPT on visit 1 (week 2), the first of 5 nutritional interventions will begin with the objective of consuming ~ 350 mg of nitrate daily from vegetables
  Arms: Intervention

SUMMARY:
Vegetables, mainly green leafy ones and some others like beets, are a rich source of nitrate. Nitrate metabolism has shown benefits to the body and there are recent studies that agree that the consumption of nitrates from vegetables can modify the oral microbiota by increasing species with nitrate-reducing capacity, which are also bacteria that are associated with oral health.

DETAILED DESCRIPTION:
Background. Periodontitis (PD) is a chronic, multifactorial and inflammatory disease caused by the imbalance resulting from the proliferation of certain pathogenic bacteria that alter the symbiotic community and cause oral dysbiosis. Non-surgical periodontal treatment (NSPT) helps to eliminate the pathogenic plaque present and it is of interest to look for adjuvant treatments that contribute to an improvement in oral health, given that, with the passage of time, a recolonization of pathogenic bacteria has been observed, as well as a relapse in patients. The oral microbiota plays a key role in the nitrate reduction process in humans, as certain bacteria reduce exogenous nitrate to nitrite, which is subsequently converted in the body to nitric oxide. Vegetables, mainly green leafy vegetables and some others such as beets, are a rich source of nitrate. Nitrate metabolism has shown benefits for the body and recent studies agree that consumption of nitrates from vegetables can positively modify the oral microbiota. Therefore, we hypothesize that the consumption of vegetables may be an adjuvant in the recovery and improve the condition of patients receiving NSPT and possibly prevent relapse.

Objective. To evaluate the effect of nitrate-rich vegetable intake on salivary levels of inflammatory molecules, nitratoreductive capacity and oral microbiota composition in patients with PD.

Material and methods. A parallel randomized clinical trial (RCT) will be conducted in 60 PD patients who are candidates for NSPT and they will be randomized into two groups. The control group will receive the NSPT and instructions to continue with their usual diet, while the intervention group, in addition to the NSPT, will receive a nutritional intervention to promote the daily consumption of vegetables rich in nitrate. The nutritional intervention will be based on the theory of the wheel of behavior change to achieve the consumption of vegetables rich in nitrate that provide ~ 350 mg of this compound. Both groups will be evaluated before and after the study: clinical, dental, and nutritional parameters. Blood samples will also be taken for blood chemistry and saliva to perform a nitratoreduction test, quantify the amount of nitrates and nitrites and determine the levels of inflammatory molecules, as well as subgingival plaque and tongue scraping, from which DNA will be extracted to be sequenced and to obtain the diversity and abundance of bacteria at the beginning, end of the RCT, 6 months and 12 months later in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and/or women from 30 to 65 years old
* Voluntary participation and signing the written informed consent
* Not receiving nutritional treatment at the time of uptake
* Availability to attend all scheduled visits
* Have an indication to receive nonsurgical periodontal treatment (NSPT)
* Interdental clinical insertion loss ≥3mm and ≥5mm in the buccal or oral area of two or more non-adjacent teeth
* Detectable depths ≥ 5mm in two or more teeth
* Radiographic evidence of periodontal bone loss

Exclusion Criteria:

* Trauma-Induced Gingival Recessions
* Cervical caries
* History of bleeding diathesis
* Pregnant or nursing women
* BMI <18.5 kg / m2
* History of any of the following self-reported diseases: type 2 diabetes mellitus, high blood pressure, kidney or liver disease, inflammatory bowel diseases, autoimmune diseases and/ or use of medications to control these diseases.
* Having or presenting a high risk of infection by tuberculosis, hepatitis B or Human Immunodeficiency Virus (HIV)
* Use of antibiotics (including antibiotic oral rinse) 6 months prior to or during the study
* Having received specialized periodontal treatment in the previous 6 months.
* Smoking habit
* Require an interpreter or not understand Spanish to attend or provide written material.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Composition of the oral microbiota | 10 weeks, 6 and 12 months
  The composition of the oral microbiota will be before and after the intervention will be evaluated in both study groups using 16S rRNA gene Illumina sequencing. For their analysis, alpha diversity will be evaluated: richness using the Chao1 index and diversity using the Shannon index; beta diversity with PCoA (principal coordinates analysis). In addition, taxonomic assignment will be performed with the DADA2 protocol at both genus and species (ASVs) level, against the SILVA database.
Evaluation of nitrate-reducing capacity | 10 weeks, 6 and 12 months
  The nitrate-reducing capacity in the mouth will be evaluated before and after the intervention in both study groups. Nitrite and nitrate levels will be quantified in saliva and in a nitrate reduction test. Test strips will be used and measured in a Merck reflectometer, which will provide the mg/L of each metabolite.
Dietary intake of nitrate | 10 weeks, 6 and 12 months
  Three 24-hour diet recall will be performed and the average nitrate intake in g/day will be evaluated. Tables reporting the average amount of nitrate in food will be used and multiplied by the reported amount of food consumed by the participant.
Periodontal chart evaluation | 10 weeks, 6 and 12 months
  Periodontal chart is a tool used by dental professionals to evaluate different parameters such as probing depth, clinical attachment level (CAL), bleeding on probing (BP), plaque or calculus (PoC), which help to identify the condition of the periodontal tissues and determine the status of the disease. The measurement of these parameters may give an indication of the extent and severity of the periodontal disease, a Hu Friedy periodontal probe is used for the evaluation, each tooth is divided into six points for study in the vestibular or lingual and palatal aspect, mesial, central and distal. A periodontist will perform the periodontal chart before and after the intervention in both study groups. The online periodontogram of the Spanish Society of Periodontology and Osseointegration (SEPA) will be used: http://sepa.es/periodontograma/index.html
Determination of salivary inflammatory molecules | 10 weeks, 6 and 12 months
  To obtain the saliva sample, the patient will be provided with a sterile 15 ml tube to deposit the accumulated saliva for 5 minutes, this time will be to obtain the largest possible amount of saliva. The saliva sample will not be stimulated (drooling or salivating). Once 3 ml are obtained, the donation will be finished. The saliva will be handled in a sterile area, 40 µl of metalloproteinase inhibitor will be added for each milliliter of saliva to avoid degradation of the molecules of interest, then it will be centrifuged at 4°C at 3,500 rpm for 10 minutes and, once the centrifugation is finished, 250 µl will be aliquoted in 1.5 ml microtubes (a total of 4 tubes) for the determination of the molecules with ELISA kit.

SECONDARY OUTCOMES:
Probing depth (PD) | 10 weeks
  The periodontal probe is inserted along the root surface of the tooth in order to measure the distance from gingival margin to pocket bottom of the periodontal pocket. The values are measured in mm, six sites per tooth, measurements are expressed as averages.
Clinical attachment level (CAL) | 10 weeks
  The clinical attachment level provides an estimation of the true periodontal support and is used for monitoring changes in periodontal support over the time.
  The "Attachment Level" for each site will be calculated based on the following formula: probing depth (mm) less gingival margin (mm) if the cemento-enamel junction (CEJ) is cover to the gingival margin. In situation where the gingival margin is apical to the CEJ, probing depth (mm) sum the distance to CEJ at gingival margin (mm). The values are measured in mm, six sites per tooth for each teeth present in the mouth, measurements are expressed as averages.
Bleeding on probing (BP) | 10 weeks
  The periodontal probe is carefully introduced to the bottom of the pocket and gently moved laterally around the tooth, six points are recorded for each tooth as bleeding present or absent, the measurements are expressed as percentage of bleeding on probing of teeth present in the mouth.
  The bleeding in each tooth is identified and the values obtained are used to average the bleeding.
Plaque or calculus (PoC) | 10 weeks
  The presence of plaque and calculus is evaluated and marked as present or absent on the periodontal chart based on 6 points on the tooth, the measurements are expressed as percentage of plaque or calculus (PoC).

CONTACTS AND LOCATIONS:
Overall Officials: Lucrecia Carrera, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Integral Dental Clinics CUCS UDG, Guadalajara, Jalisco, Mexico